CLINICAL TRIAL: NCT02111291
Title: Clinical Outcomes Associated With Enzymatic Debridement of Diabetic Foot Ulcers for Up To 12 Weeks With Clostridial Collagenase (Santyl®) Ointment
Brief Title: Santyl Applications to Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-101-09-034
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Diabetic Foot Ulcers; Diabetic Foot Wounds
Keywords: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Hydrogels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SANTYL® (Experimental)
  Interventions: Biological: Collagenase SANTYL® Ointment
- Supportive Care (Sham Comparator)
  Interventions: Biological: Hydrogel (if needed) and foam dressing

INTERVENTIONS:
Biological: Collagenase SANTYL® Ointment — Daily application directly to the ulcer bed, approximately 2 mm thick.
  Arms: SANTYL®
Biological: Hydrogel (if needed) and foam dressing — Daily application of hydrogel directly to the ulcer bed (if necessary), covered with foam dressing
  Arms: Supportive Care

SUMMARY:
The current trial examines the potential benefits of continuous 12 week treatment with Santyl, measured in terms of wound bed appearance. The visual appearance of granulation tissue will be recorded at each visit for the purpose of examining the relationship between wound bed appearance and progress towards healing. In support of this longer treatment regimen with Santyl, a recent animal study found that application of Santyl for 12 weeks was safe and well tolerated. Therefore, the present study is designed to test the hypothesis that daily treatment of diabetic foot ulcers (DFU) with Santyl for up to 12 weeks will result in more rapid development of granulation tissue than DFU treated with supportive care.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered qualified for enrollment if they meet the following criteria:

1. Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information.
2. Eighteen (18) years of age or older, of either sex, and of any race or skin type provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
3. Willing and able to make all required study visits.
4. Able to follow instructions and perform the dressing changes at home or have a caregiver who can perform the dressing changes according to the protocol.
5. Willing to use an appropriate off-loading device whenever necessary to keep weight off of any foot ulcers.
6. An ulcer present on any part of the plantar surface of the foot or plantar surface of the hallux which is 0.5 cm2 - 10 cm2 inclusive (as measured at the Screening Visit) with a duration ≥ 6 weeks but not more than 52 weeks (12 months) documented in the patient's history or by patient report of onset which requires debridement.
7. Adequate arterial blood flow as evidenced by an ankle brachial index (ABI) of > 0.70 and ≤ 1.20. If ABI > 1.2, perfusion at or near the site of the ulcer should be confirmed; the foot is warm to the touch and has palpable pulses.
8. Separation of at least 5 cm (closest ulcer edge to other closest ulcer edge) if ≥ 2 ulcers are present.
9. Diabetes mellitus (Type 1 or 2) requiring insulin or oral/injectable medications to control blood glucose levels.
10. Target ulcer is not infected based on clinical assessment.

Exclusion Criteria:

Any one (1) of the following criteria will disqualify a potential Subject from participation in the study.

1. Contraindications or hypersensitivity to the use of clostridial collagenase or hydrogel.
2. Undergoing therapy with another investigational agent within thirty (30) days of Visit 1, or planned participation overlapping with this study.
3. Bleeding disorder that would preclude sharp debridement during the study.
4. Active cellulitis of the target ulcer, lymphangitic streaking, deep tissue abscess, gangrene, or infection of muscle, tendon, joint or bone.
5. Infection with systemic toxicity or metabolic instability (e.g., fever, chills, tachycardia, hypotension, confusion, vomiting, leukocytosis, acidosis, severe hyperglycemia, azotemia).
6. A target ulcer which involves the underlying tissues of tendon, muscle, or bone.
7. Diagnosis of chronic granulomatous disease, leukocyte adhesion defects, or severe neutropenia.
8. Current treatment (at the time of the Screening Visit) with any of the following:

   * Systemic corticosteroids. If corticosteroid treatment was for ≥ 10 days, there must be a 1 week interval between discontinuation and screening.
   * Immunosuppressive agents
   * Chemotherapeutic agents
   * Antiviral agents
   * Systemic antibiotic therapy or topical antibiotic treatment of the target ulcer
9. Treatment of target ulcer with bioactive therapies within 1 month of screening:

   * Platelet-derived growth factor (e.g., Regranex)
   * Living skin equivalent (e.g., Apligraf)
   * Dermal substitute (e.g., Dermagraft, Integra, Oasis, etc.)
10. Treatment of target ulcer for any length of time with clostridial collagenase ointment (SANTYL®) if within 12 weeks prior to screening.
11. Target ulcer that failed to develop well-established granulation tissue when treated with clostridial collagenase ointment (SANTYL®) for at least 4 weeks.
12. Radiation therapy to the target lower extremity within 30 days prior to screening.
13. Medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.
14. Blood counts and blood chemistry values as follows:

    * Alanine aminotransferase (ALT) > 3x upper limit of normal
    * Aspartate aminotransferase (AST) > 3x upper limit of normal
    * Gamma Glutamyl Transferase (GGT) > 2.5x upper limit of normal
    * Serum albumin < 2.0 g/dL • Pre-albumin levels of < 10 mg/dL
    * Alkaline phosphatase > 500 U/L • Serum total bilirubin > 3.0 mg/dL
    * Serum BUN > 75 mg/dL • Serum creatinine > 4.5 mg/dL
    * HbA1c > 12% • Hemoglobin (Hgb) < 8.0 g/dL
    * WBC < 2.0 x 109/L • Absolute neutrophil count < 1.0 x 109/L
    * Platelet count < 50 x 109/L • INR > 1.5x upper limit of normal

Furthermore, prior to randomization at Visit 1, the following exclusion criteria will apply:

1. Use of excluded concomitant medications or therapies between Screening and Visit 1.
2. A clinically diagnosed infection of the target ulcer requiring treatment.
3. Muscle, tendon, or bone exposure in the target ulcer.
4. After debridement at Visit 1, the ulcer area is >12 cm2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to Well-established Granulation Tissue | 12 Weeks

SECONDARY OUTCOMES:
Adverse Event | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hebert B Slade, MD, Study Chair — Smith and Nephew Biotherapeutics
Locations (25):
- United States (22):
  - Mesa, Arizona
  - Carlsbad, California
  - Castro Valley, California
  - Fair Oaks, California
  - Fresno, California
  - Sylmar, California
  - Doral, Florida
  - Warner Robins, Georgia
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - New York, New York
  - Greenville, North Carolina
  - Reading, Pennsylvania
  - York, Pennsylvania
  - Fort Worth, Texas
  - McAllen, Texas
  - Temple, Texas
  - St. George, Utah
  - Roanoke, Virginia
  - Virginia Beach, Virginia
- Canada (3):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Montreal, Quebec